CLINICAL TRIAL: NCT06339697
Title: Short-term Effects of Bowel Preparation on Gut Microbiome in Patients Undergoing Endoscopic Colon Polypectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zhang Yanli (Other)
Responsible Party: Sponsor-Investigator, Zhang Yanli, Deputy Head of Gastroenterology, China-Japan Friendship Hospital
Organization: China-Japan Friendship Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-KY-233
Record Dates: First submitted 2024-02-28; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Colon Polyp; Cathartic Colon
Keywords: bowel preparation; gut microbiome; Cathartics
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- compounded polyethylene glycol electrolyte dispersions (Active Comparator): For patients undergoing colonoscopic polypectomy in the morning, 2-3 L should be taken the night before and 1-2 L the morning of the procedure, and for patients undergoing colonoscopy in the afternoon, divided doses should be taken on the same day.
  Interventions: Drug: different types of laxatives (compounded polyethylene glycol electrolyte dispersions and compounded sodium pico-sulfate)
- compounded sodium pico-sulfate (Active Comparator): Oral sodium picolinate/magnesium citrate (PicolaxÒ), 2 sachets, each sachet contains 0.01 g of sodium picolinate, 3.5 g of magnesium oxide, 12.0 g of citric acid, each sachet should be dissolved in 150 ml of water, sachet 1 should be taken at 7:00 p.m.-9:00 p.m. on the first day of the operation, and cite 1,500-2,000 ml of clarified fluids after the dose and before going to bed, sachet 2 should be taken 4-6 hours prior to colonoscopy, and 750 ml of clarified fluids should be taken orally before the colonoscopy. The second bag should be taken 4-6 hours before the colonoscopy and 750 ml of clarified liquid should be taken orally before the colonoscopy.
  Interventions: Drug: different types of laxatives (compounded polyethylene glycol electrolyte dispersions and compounded sodium pico-sulfate)

INTERVENTIONS:
Drug: different types of laxatives (compounded polyethylene glycol electrolyte dispersions and compounded sodium pico-sulfate) — Bowel preparation with different types of laxatives (compounded polyethylene glycol electrolytes and compounded sodium picosulfate)

SUMMARY:
To investigate the role of different types of laxatives (compounded polyethylene glycol electrolyte dispersions and compounded sodium pico-sulfate) on the composition, evolution and recovery of the gut microbiome of patients with colonic polyps undergoing bowel preparation.

DETAILED DESCRIPTION:
Good and adequate bowel preparation is essential for colonoscopy, especially in patients requiring endoscopic treatment, and the role of bowel purgatives and their safety for patients has been extensively studied. There are several laxatives available in clinical practice, the most widely used being electrolyte-supplemented polyethylene glycol (PEG) solutions, and other types of laxatives such as compound sodium picosulfate (SP) have been developed subsequently.

When a large amount of laxative passes through the intestine, many microorganisms are removed from the intestine. Thus leading to significant changes in the composition of the intestinal microbiota during intestinal cleansing. There is no consensus on how gut cleansing affects the gut microbiome.

There are no studies exploring whether there are differences in the effects of different types of laxatives on the human gut microbiome. In this study, focusing on patients diagnosed with colon polyps, the investigators explored the effects on the composition, evolution, recovery and functional pathways of the patients' gut microbiome after the use of different types of laxatives and endoscopic treatment.

ELIGIBILITY:
Inclusion Criteria:

* All colon polyps diagnosed by electronic colonoscopy
* Age above 18 years old
* Patients sign an informed consent form, agree to cooperate with the study of this project, and collect fecal specimens on time to receive follow-up visits

Exclusion Criteria:

* Patients who received antibiotics, PPIs 2 weeks before the study
* Patients who consumed probiotics or herbs 2 weeks prior to the study
* Had a colonoscopy or used diarrhea-inducing drugs or gastrointestinal stimulants 1 week prior to the study
* Gastrointestinal surgery and gastrointestinal endoscopic procedures in the 1 month prior to the study
* Bacterial or parasitic intestinal infections in the 1 month prior to the study
* Patients on long-term low-calorie diets, vegan diets, gluten-free diets and other "special" diets
* Pregnant/nursing patients
* Patients with a history of hypersensitivity to relevant medications
* Patients with contraindications to sodium picosulfate: renal insufficiency, renal transplant recipients, congestive heart failure, symptomatic ischemic heart disease within the last 6 months, cirrhosis of the liver, patients on hemodialysis or peritoneal dialysis, patients taking certain medications - renin-angiotensin blockers, diuretics, non-steroidal anti-inflammatory drugs (NSAIDs), and patients taking medications known to trigger the syndrome of inappropriate secretion of antidiuretic hormone. patients taking medications known to induce the syndrome of inappropriate antidiuretic hormone secretion (tricyclic antidepressants, selective 5-hydroxytryptamine reuptake inhibitors, multiple antipsychotics, and carbamazepine)
* Patients with contraindications to colonoscopy, such as severe hypertension, anemia, coronary artery disease, cardiopulmonary insufficiency, etc.
* Patients with contraindications to drug-induced diarrhea, such as intestinal obstruction, electrolyte disorders, or severe renal insufficiency.
* Any other reason the investigator considers inappropriate for enrollment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
gut microbiome-taxonomy | Before bowel preparation, 7 days after bowel preparation, 14 days after bowel preparation
  16s sequencing results of feces. Based on the abundance information (absolute and relative) from ZOTU and its taxonomic annotations, the total number of sequences at each taxonomic level (Kingdom, Phylum, Class, Order, Family, Genus) for each sample and its proportion of the total number of sequences were summarized.
gut microbiome-heatmap | Before bowel preparation, 7 days after bowel preparation, 14 days after bowel preparation
  Based on the species annotations and abundance information of all samples at the genus level, the genera of concern (30 genera with high default abundance rankings) and their abundance information in each sample are selected to draw heat maps. At the same time, and clustering at both the level of taxonomic information and differences between samples, one can look for patterns of aggregation of species or samples.
gut microbiome-Alpha Diversity | Before bowel preparation, 7 days after bowel preparation, 14 days after bowel preparation
  Includes both the diversity of species in the sample (Richness) and the overall evenness of the distribution of how many species make up the sample (Evenness). Indices such as Richness, Chao1, Shannon, Simpson, Dominance and Equitability are commonly used to assess the species diversity of a sample.
gut microbiome-Beta Diversity | Before bowel preparation, 7 days after bowel preparation, 14 days after bowel preparation
  Beta Diversity is a comparison of microbial community composition between samples. Bray Curtis, Weighted UniFrac and Unweighted UniFrac distances were calculated based on the ZOTUs abundance information of the samples to assess the differences in microbial community composition between samples. Based on the above distance matrix, it was analyzed by multivariate statistical methods such as Principal Component Analysis, Principal Co-ordinates AnalysisUnweighted Pair-group Method with Arithmetic Means to further from the results to explore the differences in microbial community structure in each sample and the differences in the contribution of different classifications to the samples.
gut microbiome-Functional predictions | Before bowel preparation, 7 days after bowel preparation, 14 days after bowel preparation
  In the 16S analysis, a preliminary functional spectrum prediction analysis was performed. The constructed ZOTU sequences were aligned with bacterial 16S sequence databases of known function (e.g., KEGG 16S Sequence Database, Silva SSU Database,) to obtain information on bacterial abundance in environmental samples. This abundance information is mapped directly or indirectly to the annotated microbial genomes of the KEGG databases, combined with the number of 16S rRNA genes and the abundance information of the functional genes (characterized using the KEGG Ortholog, KO), to obtain functional data on (some of the) known bacteria contained in the samples, as well as their abundance information.

SECONDARY OUTCOMES:
Age | Before bowel preparation
  Age (how old)
Gender | Before bowel preparation
  Male or female
Height | Before bowel preparation
  How many centimeters?
Weight | Before bowel preparation
  How many kilograms?
BMI | Before bowel preparation
  kg/cm2
Whether the enrollee is a smoker | Before bowel preparation
  Defined as current regular cigarette smoking
Whether the enrollee is a drinker | Before bowel preparation
  Defined as drinking of alcohol at least three times per week
Evaluation of the effectiveness of intestinal cleansing Evaluation of the effectiveness of intestinal cleansing | Within 24 hours after bowel preparation
  A Boston Rating Scale was used, with cleanliness on a 4-point scale (0-3) and a total score (0-9).
Gastrointestinal Symptom Score | Within 2 weeks after bowel preparation
  The Gastrointestinal Symptom Rating Scale (GSRS) consists of 15 questions covering 5 aspects of gastrointestinal symptoms: abdominal pain (including abdominal pain, nausea and vomiting), reflux, diarrhea (including diarrhea, loose stools, incontinence of stool, and urgency to defecate), dyspepsia (including ringing in the abdomen, abdominal distention, belching, and increased exhaustion of gas), constipation (including constipation, hard stools, and incomplete evacuation of bowel movements), with 4 answers per question. Each question provided 4 answers, and each symptom was scored from mild to severe, with scores ranging from 0 to 3. Finally, each item was summed up to give a total score, with higher scores suggesting that the patient's gastrointestinal symptoms were more severe. All the scales were filled out independently within 10-15 minutes by a uniformly trained physician who instructed the patients to review their symptoms within 1 month.
adverse event | Within 2 weeks after bowel preparation
  Any discomfort complained of by the patient

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT06339697/Prot_SAP_000.pdf